CLINICAL TRIAL: NCT07170488
Title: Post Traumatic Growth After Concussion in Women
Brief Title: Yoga and Female Concussion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: PINK Concussions (Unknown); LoveYourBrain Foundation (Unknown); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Martina Anto-Ocrah, Assistant Professor, University of Pittsburgh
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY23090017; K01NS121199 (NIH)
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Results first posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Concussion Mild
Keywords: female; women; concussion
MeSH Terms: conditions — Brain Concussion | interventions — Yoga

STUDY DESIGN:
Intervention Model Description: Because all participants will be receiving the Yoga intervention eventually (using a sequential design), allocation will be on a first come, first serve basis. After the n=15 has been reached for the Yoga, those still interested and available will be put in the wait-list control group to also receive the Yoga after the original Yoga group has finished all intervention activities.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga group (Experimental): The Yoga group were assigned to a six-week, evidence-based, light intensity Yoga and meditation curriculum developed for individuals living with TBI. The intervention is delivered online and synchronously, the program is led by experienced instructors with more than a decade of teaching experience in Yoga. Each weekly session is 75 minutes and combines gentle postures, guided breathing exercises (pranayama), Yoga nidra (deep relaxation), and meditation practices. Before each of the Yoga sessions, participants are e-mailed prerecorded tools that focused on a specific theme for the week
  Interventions: Behavioral: Yoga
- Wait List Control Group (Other): This is the wait list control group that got the Yoga intervention after data collection was completed for the Yoga group.
  Interventions: Behavioral: Yoga for wait list control

INTERVENTIONS:
Behavioral: Yoga — The LoveYourBrain (LYB) Yoga program is a six-week, evidence-based, light intensity Yoga and meditation curriculum developed for individuals living with TBI. It is delivered online and synchronously, the program is led by experienced instructors with more than a decade of teaching experience in Yoga. Each weekly session is 75 minutes and combines gentle postures, guided breathing exercises (pranayama), Yoga nidra (deep relaxation), and meditation practices. Before each of the Yoga sessions, participants are e-mailed prerecorded tools that focused on a specific theme for the week (resilience, mindfulness etc.)
  Other Names: LoveYourBrain Yoga
  Arms: Yoga group
Behavioral: Yoga for wait list control — After the active Yoga group received the intervention, the wait list control was then assigned to the intervention.
  Arms: Wait List Control Group

SUMMARY:
Most research on the impact of mild Traumatic Brain Injury/Concussions have been deficit-based and focused on the impairments induced by the injury. Research shows that trauma doesn't always have negative effects. While some people suffer, others may experience positive psychological changes. This is known as posttraumatic growth (PTG), which refers to the positive changes that can come from struggling with a life-changing event. In this study, the investigators explore if pilot yoga intervention improves PTG scores for women who have had concussions.

DETAILED DESCRIPTION:
The investigators will be collaborating with the Pink Concussion network on this endeavor to recruit study participants who are residents of United States. PINK is an online support network for women with concussion symptoms lasting ≥1 month. PINK participants will be recruited online using an IRB approved consent form that will be on the study's landing page. Upon clicking the survey invitation link, potential survey takers will be brought to the very first page of the survey which will be the IRB-approved consent page. This will list the risks, benefits, incentives, and overall research processes. The consent will also state that the research is no greater than minimal risk and involves procedures for which written consent is normally not required outside of the research context. After reviewing the approved information sheet, participants will be prompted to consent yes in order to move on to the survey body. Those who do not consent will be sent to a "Thank you page" and not continue. Those who do so, will begin the survey. All survey questions will be voluntary and responses will be de-identified and analyzed in aggregate to ensure anonymity.

The Yoga intervention will be administered by LoveYourBrain Yoga, a US-based global non-profit organization that aims to improves the quality of life of people affected by traumatic brain injury through Yoga and meditation, education and other brain-health initiatives.

Thirty PINK participants will be randomly selected to participate in the LYB Yoga intervention. The Yoga sessions will be virtual and study participants will be able to complete these sessions at home. The session will not be recorded. They will be free of cost for the study participants. Yoga that will be taught is a simple form of exercise that is tailored to people with a history of TBI. The movements are slow and study participants will have the choice to participate up to their comfort level.The role of LoveYourBrain will be to administer the yoga intervention and will not be engaged in the research study.

The investigators will administer the Post-Traumatic Growth surveys again at 7 weeks and 30 days to 15 Yoga and 15 Wait list controls. The 15 Yoga participants will also do the post-yoga assessments at 7 weeks (1 week post-yoga). The 15 Wait list controls will do the LYB program after the 30-day PTG surveys have been completed. The 15 Wait list controls will receive a follow up survey, 1 week after the completion of the LYB program. The intervention group participants who have attended 3 or more LYB yoga sessions will also receive a week-20 follow up survey. Total evaluations will be at 1 week, 5 weeks and 20 weeks post-yoga

Because all participants will be receiving the Yoga intervention eventually (using a sequential design), allocation will be on a first come, first serve basis. After the n=15 has been reached for the Yoga, those still interested and available will be put in the wait-list control group to also receive the Yoga after the original Yoga group has finished all intervention activities.

ELIGIBILITY:
Inclusion Criteria for ALL PINK participants (STEP 1):

* 18 years of age or older
* Assigned female at birth
* Belongs to PINK Concussion Facebook group from as a concussion survivor
* Should be a resident of United States

Exclusion Criteria:

• Does not consent to study

To be included in YOGA intervention from STEP 1, they should:

1. Have low PTG (PGI-X score <75)
2. Be inexperienced/novice yoga users
3. Not be receiving rehab services

Exclusion Criteria:

* Does not consent to study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-11-10 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-04-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, DGIM, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Data will be analyzed in aggregate and there is no plans to share participant data individually. We must protect their identity and ensure data anonymity and confidentiality. This is particularly important given the small sample sizes. Upon reasonable request from the PI, Dr. Anto-Ocrah, the data will be shared in aggregate.

REFERENCES:
- [Background] Donnelly KZ, Baker K, Pierce R, St Ivany AR, Barr PJ, Bruce ML. A retrospective study on the acceptability, feasibility, and effectiveness of LoveYourBrain Yoga for people with traumatic brain injury and caregivers. Disabil Rehabil. 2021 Jun;43(12):1764-1775. doi: 10.1080/09638288.2019.1672109. Epub 2019 Oct 2. PMID 31577456
- [Background] Callahan CE, Beisecker L, Zeller S, Donnelly KZ. LoveYourBrain Mindset: Feasibility, Acceptability, Usability, and Effectiveness of an Online Yoga, Mindfulness, and Psychoeducation Intervention for People with Traumatic Brain Injury. Brain Inj. 2023 Apr 16;37(5):373-382. doi: 10.1080/02699052.2023.2168062. Epub 2023 Jan 24. PMID 36692090
- [Background] Donnelly KZ, Linnea K, Grant DA, Lichtenstein J. The feasibility and impact of a yoga pilot programme on the quality-of-life of adults with acquired brain injury. Brain Inj. 2017;31(2):208-214. doi: 10.1080/02699052.2016.1225988. Epub 2016 Dec 12. PMID 27936953
- See also: PINK Concussions. PINK concussions: Female brain injury from sports, violence, military service — https://www.pinkconcussions.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Yoga Group | Wait List Control Group
Started | 12 | 15
Completed | 5 | 11
Not Completed | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Yoga Group | Wait List Control Group | Total
Number analyzed (Participants) | 12 | 15 | 27
Age, Continuous [Mean (Full Range); unit: Years] | 46.6 [22 to 67] | 35.8 [24 to 53] | 40.8 [22 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10 | 10 | 20
  Black/AA | 1 | 5 | 6
  Hispanic | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Post Traumatic Growth
Description: Post Traumatic Growth Inventory (PTGI-X). Scores range from 0-125, with higher scores indicating greater post traumatic growth. Scores ≥75 is used as cutoff for moderate to high PTG; and scores <75 are deemed low PTG
Time Frame: Baseline (at enrollment), 1 week post-yoga (Week 7) and 4 weeks post-yoga (Week 10), and Week 19 (after the wait-list control group had completed their yoga sessions)
Population: Response rate at week 19 was much lower than earlier timepoints, leading to a smaller size. We completed the analyses for those without missing data.
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Yoga Group | Wait List Control Group
Number analyzed (Participants) | 5 | 11
Score on a scale
  Baseline (at enrollment) | 41.7 [14 to 59] | 57.8 [40 to 73]
  1 week post-yoga (Week 7) | 40.4 [1 to 61] | 60.7 [13 to 120]
  4 weeks post-yoga (Week 10) | 32.5 [0 to 39] | 11 [3 to 113]
  Week 19 (after the wait-list control group had completed their yoga sessions): number analyzed (Participants) | 4 | 4
  Week 19 (after the wait-list control group had completed their yoga sessions) | 37.6 [0 to 48] | 71.5 [22 to 112]

2. Secondary Outcome: Female Sexual Function Index-6 (FSFI-6)
Description: To assess intimacy/relationships after brain injury. Consists of 6 questions related to sexual activity within the 4 weeks prior to the examination and includes sexual desire, sexual arousal, lubrication, orgasm, satisfaction, and pain. Scoring is based on Likert scoring from 0-5. Total scores range from 2-30 with lower scores corresponding to worse sexual functioning.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Yoga Group | Wait List Control Group
Number analyzed (Participants) | 5 | 11
Score on a scale
  Baseline (at enrollment) | 11 [0 to 26] | 19.15 [0 to 28]
  1 week post-yoga (Week 7) | 17.5 [0 to 27] | 20.18 [8 to 27]
  4 weeks post-yoga (Week 10) | 16.75 [0 to 28] | 19.27 [8 to 29]
  Week 19 (after the wait-list control group had completed their yoga sessions): number analyzed (Participants) | 4 | 4
  Week 19 (after the wait-list control group had completed their yoga sessions) | 12.2 [0 to 19] | 23 [19 to 27]

3. Other Pre Specified Outcome: Rivermead Post-Concussion Questionnaire
Description: The investigators will use the Rivermead Post-Concussion Questionnaire to evaluate prevalence of persistent Post-concussion Symptoms among study participants. The RPQ is a 16-item self-report measure of the presence and severity of the 16 most commonly reported post-concussive symptoms observed in the literature. Values for each of the 16 items are ranked on a five-point scale (0 = not experienced at all, 4 = severe problem). Scores on the RPQ range from 0 to 64, with higher scores suggestive of greater PCS burden.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Yoga Group | Wait List Control Group
Number analyzed (Participants) | 5 | 11
Score on a scale
  Baseline (at enrollment) | 35.4 [28 to 45] | 26 [1 to 44]
  1 week post-yoga (Week 7) | 35.7 [26 to 46] | 25 [1 to 37]
  4 weeks post-yoga (Week 10) | 36 [24 to 52] | 11 [0 to 40]
  Week 19 (after the wait-list control group had completed their yoga sessions): number analyzed (Participants) | 4 | 4
  Week 19 (after the wait-list control group had completed their yoga sessions) | 34.3 [24 to 48] | 18.3 [1 to 27]

4. Other Pre Specified Outcome: Anxiety
Description: The investigators will use the General Anxiety Disorder (GAD-7) to evaluate prevalence of anxiety post-concussion using this brief 9-item screener. Participants respond to how often they have been bothered by symptoms, from 0 (not at all) to 3 (nearly every day).GAD-7 total score for the seven items ranges from 0 to 21, with higher scores suggestive of greater anxiety.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Yoga Group | Wait List Control Group
Number analyzed (Participants) | 5 | 11
Score on a scale
  Baseline (at enrollment) | 7.7 [1 to 9] | 7.3 [3 to 11]
  1 week post-yoga (Week 7) | 3.8 [1 to 8] | 4.8 [1 to 12]
  4 weeks post-yoga (Week 10) | 6.4 [0 to 12] | 6.3 [1 to 15]
  Week 19 (after the wait-list control group had completed their yoga sessions): number analyzed (Participants) | 4 | 4
  Week 19 (after the wait-list control group had completed their yoga sessions) | 8.3 [2 to 13] | 8 [2 to 11]

5. Other Pre Specified Outcome: Depression
Description: The investigators will use the Patient Health Questionnaire (PHQ-9) to evaluate prevalence of depression post-concussion among study participants. The Patient Health Questionnaire (PHQ-9) is a 9-item screener to assess the frequency of depressed mood/anhedonia over the past two weeks. Participants respond to how often they have been bothered by symptoms, from 0 (not at all) to 3 (nearly every day). Scores range from 0-27, with higher scores suggestive of greater depression.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Yoga Group | Wait List Control Group
Number analyzed (Participants) | 5 | 11
Score on a scale
  Baseline (at enrollment) | 9.5 [5 to 16] | 9.2 [1 to 17]
  1 week post-yoga (Week 7) | 7.6 [4 to 17] | 7.4 [2 to 19]
  4 weeks post-yoga (Week 10) | 9 [3 to 16] | 8.2 [0 to 16]
  Week 19 (after the wait-list control group had completed their yoga sessions): number analyzed (Participants) | 4 | 4
  Week 19 (after the wait-list control group had completed their yoga sessions) | 9.6 [3 to 17] | 8.8 [0 to 14]

6. Other Pre Specified Outcome: Post Traumatic Stress Disorder (PTSD)
Description: The investigators will use the PTSD Checklist for The Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM-V) (PCL-5) to evaluate prevalence of PTSD among study participants. This is a well-validated 20-item scale that assesses symptoms mirrored from the diagnostic criteria for PTSD in the DSM-V. Participants rate the extent that symptoms have bothered them in the past month on a 5-point scale from 0-4, with total scores ranging from 0-80 and higher scores indicating greater symptom severity.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Yoga Group | Wait List Control Group
Number analyzed (Participants) | 5 | 11
Score on a scale
  Baseline (at enrollment) | 28.2 [5 to 68] | 26.7 [4 to 60]
  1 week post-yoga (Week 7) | 19.2 [2 to 47] | 22.2 [0 to 51]
  4 weeks post-yoga (Week 10) | 23.4 [3 to 52] | 26.2 [2 to 60]
  Week 19 (after the wait-list control group had completed their yoga sessions): number analyzed (Participants) | 4 | 4
  Week 19 (after the wait-list control group had completed their yoga sessions) | 28.3 [2 to 57] | 28.5 [0 to 41]

7. Secondary Outcome: Resilience
Description: Resilience will be measured using the 25-item Resilience Scale. Range of scores: 25 - 175; higher scores indicating greater resilience
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Yoga Group | Wait List Control Group
Number analyzed (Participants) | 5 | 11
Score on a scale
  Baseline (at enrollment) | 133.6 [100 to 160] | 134.9 [107 to 154]
  1 week post-yoga (Week 7) | 133.1 [102 to 158] | 142.4 [117 to 169]
  4 weeks post-yoga (Week 10) | 133.9 [109 to 149] | 140.2 [118 to 157]
  Week 19 (after the wait-list control group had completed their yoga sessions): number analyzed (Participants) | 4 | 4
  Week 19 (after the wait-list control group had completed their yoga sessions) | 127.3 [106 to 131] | 143.3 [124 to 154]

8. Secondary Outcome: Flourishing
Description: This 12- item scale will be used to understand overall wellbeing before and after the intervention. The score is obtained by summing the scores from the twelve questions in all six domains and results in a score from 0 - 120. Scores are on a scale of 0-10. Higher scores are indicative of greater flourishing.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Yoga Group | Wait List Control Group
Number analyzed (Participants) | 5 | 11
Score on a scale
  Baseline (at enrollment) | 72.3 [32 to 100] | 84.1 [63 to 103]
  1 week post-yoga (Week 7) | 75.3 [36 to 94] | 59 [59 to 107]
  4 weeks post-yoga (Week 10) | 73.8 [56 to 88] | 90.5 [74 to 110]
  Week 19 (after the wait-list control group had completed their yoga sessions): number analyzed (Participants) | 4 | 4
  Week 19 (after the wait-list control group had completed their yoga sessions) | 68.7 [43 to 79] | 92.5 [72 to 105]

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 20 weeks.
Arm/Group | Yoga Group | Wait List Control Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/15
Other Adverse Events (participants affected / at risk) | 0/12 | 0/15

LIMITATIONS AND CAVEATS:
This was a quasi-experimental feasibility pilot study with a targeted sample size of 30, and 16 completed (5 Yoga, 11 controls). The study is not sufficiently powered for statistical tests of significance of the primary and secondary outcome measures. Results may inform larger trials.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-06): https://cdn.clinicaltrials.gov/large-docs/88/NCT07170488/Prot_SAP_000.pdf